CLINICAL TRIAL: NCT04470284
Title: Self-Monitoring of and Feed-back Using APP. in TReatment of UnconTroled Blood Pressure (SMART-BP)
Brief Title: Mobile App for BP Control
Acronym: SMART-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Dong-Ju Choi, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART-BP
Record Dates: First submitted 2020-07-06; First posted 2020-07-14 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMBP_only (Active Comparator): Standard treatment with SMBP
  Interventions: Other: Standard SMBP
- SMBP_mobile_app (Experimental): SMBP with mobile App based feed-back algorithm
  Interventions: Other: Mobile Application

INTERVENTIONS:
Other: Mobile Application — SMBP with mobile App based feed-back algorithm. The App based feed-back algorithm will remind the patients of taking drug to improve BP control and drug compliance.
  Arms: SMBP_mobile_app
Other: Standard SMBP — Standard treatment (SMBP-alone)
  Arms: SMBP_only

SUMMARY:
SMART-BP is a randomized, controlled study in which hypertensive patients are allocated to self monitoring of blood pressure monitoring (SMBP) only group or SMBP with mobile App based feed-back algorithm (SMBP-App) group. The App based feed-back algorithm will provide the patients with instruction in response to the measured BP value, e.g. remind of taking drug, if high blood pressure is detected.

The primary outcomes are mean systolic BP change and drug compliance at 24-weeks. Secondary endpoints include mean diastolic BP change at 12-week, mean systolic and diastolic BP change at 12 and 24 weeks, and drug compliance.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, open-label, multicenter trial to evaluate the efficacy of SMBP with mobile health application (SMBP-App) compared with SMBP alone.

Patients with hypertension will be randomly assigned to SMBP-App (intervention) and SMBP along (control) groups. In SMBP group the patients perform home blood pressure measurement and usual care. In SMBP-App group the patients perform home blood pressure and receive extra alarm and instructions from the mobile application in response to the obtained blood pressure value.

The aim of this study is to evaluate whether SMBP-App is superior to SMBP alone in terms of blood pressure reduction and improved drug compliance in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with essential hypertension aged 19 years and above.
2. Patients with essential hypertension who are taking one or more antihypertensive drugs.
3. Patients whose average systolic and diastolic BP measured 3 times on the reference arm in the sitting position during Visit 1 is greater than 140 mmHg and 90 mmHg, respectively.
4. Patients voluntarily consent to participate in this clinical trial
5. Patients who can use a smartphone

Exclusion Criteria:

1. Patients with a history of secondary hypertension or suspected secondary hypertension, including coarctation of the aorta, primary hyperaldosteronism, renal artery stenosis, Cushing's syndrome, pheochromocytoma, and polycystic kidney disease.
2. Patients with a mean systolic BP ≥ 200 mmHg or diastolic BP ≥ 110 mmHg at the screening visit.
3. Patients with ≥ 20 mmHg difference between the highest and the lowest sitting systolic BP or ≥ 10 mmHg difference between highest and lowest diastolic BP, which is confirmed by triplicate measurements from the reference arm at screening.
4. Patients with uncontrolled diabetes (HbA1c ≥ 9.0%).
5. Patients who have been continuously taking other medications such as systemic steroids, thyroid hormones, oral contraceptives (except for menopausal hormone replacement therapy), psychiatric drugs, non-steroidal anti-inflammatory drugs, sympathetic drugs, and immune suppressants, which have the potential to affect BP.
6. Patients with symptomatic orthostatic hypotension.
7. Patients with a history of malignant tumors, including leukemia and lymphoma, within the past 5 years.
8. Patients with a history of autoimmune diseases, such as rheumatoid arthritis and systemic lupus erythematosus.
9. Patients with clinically significant kidney and liver diseases, such as those on dialysis, liver cirrhosis, biliary obstruction, and hepatic failure, or those who show the following findings during the screening visit:

   * Alanine transaminase or aspartate transaminase level is at least 3 times higher than the normal upper limit;
   * Total bilirubin level is more than twice the normal upper limit;
   * Blood urea nitrogen level is more than twice the normal upper limit;
   * Alkaline phosphatase level is more than twice the normal upper limit;
   * Creatinine clearance level is less than 10 mL/min.
10. Patients with a history of the following diseases in the past 6 months, which are determined to be clinically significant by the investigator:

    * Heart failure (NYHA class III and IV), ischemic heart diseases (coronary artery diseases, such as angina pectoris and myocardial infarction), peripheral vascular diseases, hemodynamically significant valve stenosis, and arrhythmia.
    * Severe cerebrovascular events, including stroke, cerebral infarction, and cerebral hemorrhage.
11. Patients with shock.
12. Patients with a history of alcohol or drug abuse.
13. Patients with potential pregnancy or breastfeeding.
14. Patients who will be judged as both legally and psychologically inadequate to participate in the clinical study by the investigator.
15. Patients who have participated in clinical studies with other investigational drug products within 4 weeks prior to screening.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
mean home systolic BP change | 24 weeks
  mean home systolic BP change from baseline to 24 weeks (Visit 2)
Drug adherence | 24 weeks
  Drug adherence using pill count

SECONDARY OUTCOMES:
Diastolic BP change | 12 weeks and 24 week
  mean home diastolic BP change from baseline
office BP change | 12 weeks and 24 week
  office systolic or diastolic BP change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ju Choi, MD, PhD, Study Chair — Seoul National Univeristy Bundang Hospital
Locations (5):
- South Korea (5):
  - Korea Univ. Guro Hospital, Seoul, Guro
  - Hallym University Sacred Heart Hospital, Anyang
  - Seoul National University Bundang Hospital, Seongnam
  - Heart Vascular Stroke Institute, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Kyung Hee University Hospital, Seoul

REFERENCES:
- [Derived] Yoon M, Hur T, Park SJ, Jo SH, Kim EJ, Kim SJ, Hussain M, Hua CH, Lee S, Choi DJ. Self-Monitoring of Blood Pressure and Feedback via Mobile App in Treatment of Uncontrolled Hypertension: The SMART-BP Randomized Clinical Trial. Mayo Clin Proc. 2025 May;100(5):840-853. doi: 10.1016/j.mayocp.2024.09.018. Epub 2025 Mar 5. PMID 40047759
- [Derived] Choi DJ, Park JJ, Yoon M, Park SJ, Jo SH, Kim EJ, Kim SJ, Lee S. Self-Monitoring of Blood Pressure and Feed-back Using APP in TReatment of UnconTrolled Hypertension (SMART-BP): A Randomized Clinical Trial. Korean Circ J. 2022 Oct;52(10):785-794. doi: 10.4070/kcj.2022.0133. PMID 36217600